CLINICAL TRIAL: NCT01312675
Title: Randomized, Multi-Centre, Controlled Clinical Study on Effect of the Selective Adsorption System for Removal of Bacterial Toxins (S.A.F.E.BT) Therapy on Disease Severity and Inflammation in Mechanically-Ventilated Subjects Due to Severe Sepsis
Brief Title: S.A.F.E.BT System Extracorporeal Treatment With DIAPACT CRRT
Acronym: SAFEbt
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped for operational futility. Due to very small numbers of subjects, insufficient data was available for results to provide meaningful conclusions.
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA-I-H-0903
Record Dates: First submitted 2011-03-08; First posted 2011-03-11 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Severe Sepsis
Keywords: severe sepsis; mechanical ventilation
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): S.A.F.E.BT plus Standard of Care therapy
  Interventions: Device: S.A.F.E.BT
- Group B (No Intervention): Standard of Care therapy alone

INTERVENTIONS:
Device: S.A.F.E.BT — Five (5) S.A.F.E.BT treatments within a 7 day treatment period.
  Arms: Group A

SUMMARY:
The purpose of this study is to determine if Selective Adsorption System for Removal of Bacterial Toxins (S.A.F.E.BT) therapy is effective in the treatment of severe sepsis.

DETAILED DESCRIPTION:
Is extracorporeal treatment effective in the treatment of sepsis

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of Sepsis
* Mechanical ventilation due to acute pulmonary dysfunction
* One additional (second) acute sepsis-related organ dysfunction

Exclusion Criteria

* Pregnant women and nursing mothers
* Conditions or medications associated with an increased risk of bleeding/complications from anticoagulation
* Previous episode of sepsis during this hospitalization
* PaO2/FiO2 ratio < 300
* Severe granulocytopenia (leukocytes <500 / μl)
* Acute hepatic diseases or severe liver failure or cirrhosis
* Chronic cardiovascular disease precluding extracorporeal treatment
* Human immunodeficiency virus complicated by AIDS defining illness
* Evidence of active bleeding - uncontrolled hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wilkins, MBChB FRCA, Study Director — BBraun Inc
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sequential Organ Failure Assessment (SOFA) Score (a.k.a. Sepsis-related Organ Failure Assessment)
Description: The primary outcome measure is the average of all changes in daily SOFA scores from baseline through Day 8.
  The SOFA score indicates quantitatively, and as objectively as possible, the degree of organ dysfunction/failure by describing a sequence of complications in the critically ill. SOFA score consists of classifications for six (6) organ functions: Respiratory, Cardiovascular, Coagulation, CNS, Liver, and Renal. Each function is assigned a value from 0 (normal organ function) to 4 (most abnormal organ function).
  Each subject's 6 organ function SOFA scores are summed to become a single daily SOFA score (total score range: 0-24, where 24 is the maximum score associated with the most abnormal function and worst outcomes). A higher SOFA score on Day 2 compared to Day 1 indicates more abnormal organ functions and a worsening physical condition.
Time Frame: Baseline through Day 8
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 9 | 7
scores on a scale
  Screening | 7.4 (2.70) | 11.9 (3.24)
  Day 1 / Baseline | 6.9 (2.57) | 11.9 (2.41)
  Day 2 | 6.9 (2.09) | 11.4 (3.10)
  Day 3: number analyzed (Participants) | 8 | 7
  Day 3 | 6.1 (2.10) | 10.4 (3.41)
  Day 4: number analyzed (Participants) | 8 | 7
  Day 4 | 6.6 (2.83) | 9.0 (3.61)
  Day 5: number analyzed (Participants) | 7 | 7
  Day 5 | 6.9 (2.97) | 7.0 (4.08)
  Day 6: number analyzed (Participants) | 7 | 7
  Day 6 | 5.6 (3.55) | 7.1 (2.85)
  Day 7: number analyzed (Participants) | 7 | 7
  Day 7 | 5.1 (3.93) | 8.1 (2.91)
  Day 8: number analyzed (Participants) | 7 | 7
  Day 8 | 4.3 (2.81) | 7.7 (1.98)

ADVERSE EVENTS:
Time Frame: 28 days per subject.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 1/9 | 1/7
Serious Adverse Events (participants affected / at risk) | 2/9 | 5/7
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=9) | Group B (N=7)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (4)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=9) | Group B (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Abdonimal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gi haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Impaired Healing (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 0 (0) | 1 (1) — Administration Site Condition
Pain (General disorders) | 1 (2) | 1 (6) — Administration Site Condition
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Brucellosis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphate increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Carbon dioxide increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (8) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (5) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (8) | 1 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (7) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (6) | 1 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Skin operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study did not reach the target number of participants needed to achieve target power and statistically reliable results leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study sites are able to publish on their own data if Sponsor does not publish a multi-center study paper within 18 months after trial completion.

Sites agree to submit any proposed publication, presentation or other public disclosure to Sponsor for review at least 30 days prior to submitting to a publisher or other 3rd party. Within 30 days of receipt, Sponsor shall advise removal of any confidential information or which may impair Sponsor's ability to obtain patent protection.